CLINICAL TRIAL: NCT00064844
Title: Combination Nicotine Replacement for Alcoholic Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAACOO11197-05; R01AA011197 (NIH)
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Smoking; Alcoholism
Keywords: Smoking; Alcoholism
MeSH Terms: conditions — Smoking; Alcoholism | interventions — Cognitive Behavioral Therapy; Ethanol; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine patch plus placebo gum (Placebo Comparator): Subjects in both arms were instructed to use one 21-mg (Nicoderm CQ®) nicotine patch daily for 8 weeks followed by one 14-mg patch daily for 2 weeks, then followed by one 7-mg patch daily for 2 weeks, for a total of 12 weeks of nicotine patch therapy. Placebo gum was given for ad libitum use, with encouragement to use at least six pieces per day, up to a maximum of 20 pieces per day. The placebo gum (manufactured by Fertin Pharma A/S, Vejle, Denmark) contained 2.6% cayenne pepper to simulate the taste of nicotine. Use of the gum was encouraged for 24 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy for alcohol and smoking cessation; Drug: Nicoderm CQ nicotine patch; Drug: Placebo gum
- Nicotine patch plus active gum (Active Comparator): Subjects in both arms were instructed to use one 21-mg (Nicoderm CQ®) nicotine patch daily for 8 weeks followed by one 14-mg patch daily for 2 weeks, then followed by one 7-mg patch daily for 2 weeks, for a total of 12 weeks of nicotine patch therapy. Nicotine gum (2 mg uncoated mint Nicorette®) was given for ad libitum use, with encouragement to use at least six pieces per day, up to a maximum of 20 pieces per day. Use of the gum was encouraged for 24 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy for alcohol and smoking cessation; Drug: Nicoderm CQ nicotine patch; Drug: Nicotine gum - Nicorette®

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for alcohol and smoking cessation — Individual 60-minute treatment sessions were scheduled weekly for the first 3 months, then monthly for the next 3 months for a total of 16 sessions. Alcohol treatment was based on the cognitive behavioral therapy manual developed for Project MATCH, with approximately 40-45 minutes of each session devoted to alcohol treatment. Components of this intervention included identifying alcohol antecedents, coping with alcohol urges, managing thoughts about alcohol, problem solving, drink refusal skills, planning for emergencies, communication and assertiveness training and enhancing social support networks for alcohol abstinence. The smoking cessation intervention was delivered in the same sessions as the alcohol treatment, with approximately 15-20 minutes of each session devoted to smoking cessation. Treatment employed behavioral elements that have been supported empirically according to the USDHHS smoking cessation practice guideline.
Drug: Nicoderm CQ nicotine patch — Subjects in both arms were instructed to use one 21-mg (Nicoderm CQ®) nicotine patch daily for 8 weeks followed by one 14-mg patch daily for 2 weeks, then followed by one 7-mg patch daily for 2 weeks, for a total of 12 weeks of nicotine patch therapy.
Drug: Placebo gum — Placebo gum was given for ad libitum use, with encouragement to use at least six pieces per day, up to a maximum of 20 pieces per day. The placebo gum (manufactured by Fertin Pharma A/S, Vejle, Denmark) contained 2.6% cayenne pepper to simulate the taste of nicotine. Use of the gum was encouraged for 24 weeks.
  Arms: Nicotine patch plus placebo gum
Drug: Nicotine gum - Nicorette® — Nicotine gum (2 mg uncoated mint Nicorette®) was given for ad libitum use, with encouragement to use at least six pieces per day, up to a maximum of 20 pieces per day. Use of the gum was encouraged for 24 weeks.
  Arms: Nicotine patch plus active gum

SUMMARY:
The overall objective of the study is to develop recommendations for treatment programs to help alcoholic smokers to stop smoking. A sample of 175 alcohol dependent cigarette smokers will be recruited from the community and treated in a 6-month outpatient alcohol and tobacco treatment program. The 175 patients will be divided into two groups. One group will receive an active nicotine patch and active nicotine gum. The other group will receive an active nicotine patch and placebo nicotine gum. Followup assessments will be conducted for 1-year from the beginning of treatment.

ELIGIBILITY:
Inclusion criteria:

* Males and females at least 18 years old.
* English speaking.
* Meets criteria for alcohol dependence or alcohol abuse.
* Must complete an alcohol detoxification program prior to entering the study.
* Currently smoking 15 or more cigarettes per day and have at least a 3 year history of smoking.
* Have a current desire to stop smoking and stop drinking.
* Willing to complete followup assessments up to 12 months after treatment.
* Willing to provide names of 2 people who can help locate the subject at followup and the name of one person who can verify information about alcohol and tobacco use.
* One person per household.

Exclusion Criteria:

* Allergy to nicotine patch or nicotine gum.
* Weigh less than 100 pounds.
* Use other nicotine products, such as cigars, pipes or smokeless tobacco.
* Severe skin disorder.
* Active peptic ulcer.
* Active joint disease.
* Heart attack within 3 months prior to entering the study.
* Pregnant or breastfeeding female who are not on birth control.
* Currently taking medication to treat alcoholism or smoking, such as naltrexone, disulfiram or bupropion.
* Poor vision or hearing that would interfere with using a cell phone.
* Lack of transportation to the treatment site or live at least one hour from the treatment site.
* Homeless.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2002-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Cooney, PhD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, Newington, Connecticut, United States

REFERENCES:
- [Background] Cooney NL, Cooney JL, Perry BL, Carbone M, Cohen EH, Steinberg HR, Pilkey DT, Sevarino K, Oncken CA, Litt MD. Smoking cessation during alcohol treatment: a randomized trial of combination nicotine patch plus nicotine gum. Addiction. 2009 Sep;104(9):1588-96. doi: 10.1111/j.1360-0443.2009.02624.x. Epub 2009 Jun 22. PMID 19549054
- [Background] Holt LJ, Litt MD, Cooney NL. Prospective analysis of early lapse to drinking and smoking among individuals in concurrent alcohol and tobacco treatment. Psychol Addict Behav. 2012 Sep;26(3):561-72. doi: 10.1037/a0026039. Epub 2011 Oct 24. PMID 22023022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 96 men and women were randomized to treatment at the Newington and West Haven campuses of the Veterans Affairs (VA) Connecticut Healthcare System.
Period: Overall Study
Arm/Group | Nicotine Patch Plus Active Gum | Nicotine Patch Plus Placebo Gum
Started | 45 | 51
2 Week Follow-up | 45 | 51
3 Month Follow-up | 40 | 47
6 Month Follow-up | 39 | 40
12 Month Follow-up | 37 | 32
Completed | 37 | 32
Not Completed | 8 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch Plus Active Gum | Nicotine Patch Plus Placebo Gum | Total
Number analyzed (Participants) | 45 | 51 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.2) | 44.8 (10.1) | 44.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 32 | 37 | 69
Region of Enrollment [Number; unit: participants]
  United States | 45 | 51 | 96

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Smoking Abstinence
Description: Percentage of participants with prolonged carbon monoxide verified smoking abstinence
Time Frame: 6 months after smoking quit date
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Nicotine Patch Plus Active Gum | Nicotine Patch Plus Placebo Gum
Number analyzed (Participants) | 39 | 40
percentage of participants abstinent | 20 | 12

2. Primary Outcome: 12 Month Smoking Abstinence
Description: Percentage of participants with prolonged carbon monoxide verified smoking abstinence
Time Frame: 12 months after smoking quit date
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Nicotine Patch Plus Active Gum | Nicotine Patch Plus Placebo Gum
Number analyzed (Participants) | 37 | 32
percentage of participants abstinent | 13 | 0
Statistical Analysis 1: Comparison: Nicotine Patch Plus Active Gum vs Nicotine Patch Plus Placebo Gum; Test type: Superiority or Other; p < 0.01, Chi-squared; df = 1, N = 96; chi square = 7.25

ADVERSE EVENTS:
Arm/Group | Nicotine Patch Plus Active Gum | Nicotine Patch Plus Placebo Gum
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/51
Other Adverse Events (participants affected / at risk) | 1/45 | 7/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch Plus Active Gum (N=45) | Nicotine Patch Plus Placebo Gum (N=51)
bleeding gums (General disorders) | 1 (1) | 7 (7)
jaw ache (General disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes